CLINICAL TRIAL: NCT03891316
Title: Human Biomonitoring of Operating Room Personnel With Occupational Exposure to the Volatile Anaesthetic Sevoflurane
Brief Title: Sevoflurane Human Biomonitoring in Operating Room Personnel
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: PV5820
Record Dates: First submitted 2019-03-10; First posted 2019-03-27 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Occupational Exposure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urinary Samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Anaesthesiologists balanced: Anaesthesiologists performing balanced anaesthesia with sevoflurane.
  Interventions: Diagnostic Test: HFIP and Sevoflurane are measured after 3 consecutive days of work.
- Anaesthesiologists TIVA: Anaesthesiologists performing only total intravenous anaesthesia.
  Interventions: Diagnostic Test: HFIP and Sevoflurane are measured after 3 consecutive days of work.
- Surgeons: Surgeons working in the operating room while anaesthesia of the patients is randomly maintained with sevoflurane or propofol.
  Interventions: Diagnostic Test: HFIP and Sevoflurane are measured after 3 consecutive days of work.
- Anaesthesiologists PACU: Anaesthesiologists working in the postoperative care unit.
  Interventions: Diagnostic Test: HFIP and Sevoflurane are measured after 3 consecutive days of work.
- Anaesthesiologists outside the operating room: Anaesthesiologists working outside of the operating room, for example pain service or anaesthesiological walk-in clinic
  Interventions: Diagnostic Test: HFIP and Sevoflurane are measured after 3 consecutive days of work.
- Physicians not exposed: Physicians not having contact with patients on wards/outpatient clinics after exposure with sevoflurane
  Interventions: Diagnostic Test: HFIP and Sevoflurane are measured after 3 consecutive days of work.
- Patients: Patients having undergone sevoflurane anesthesia for elective surgery
  Interventions: Diagnostic Test: HFIP and Sevoflurane are measured after 3 consecutive days of work.

INTERVENTIONS:
Diagnostic Test: HFIP and Sevoflurane are measured after 3 consecutive days of work. — Concentration of hexafluoroisopropanol and Sevoflurane are measured in urine by gas chromatography

SUMMARY:
Sevoflurane is a widely used volatile agent for induction and maintenance of anaesthesia. The administration of sevoflurane involves the risk of occupational exposure. Possible negative implications of chronic occupational exposure to sevoflurane are not completely refuted. In Germany no maximum workplace concentration for sevoflurane is defined. This study aims to find out if working conditions of physicians and different anaesthesia techniques effect the extent of occupational exposure to sevoflurane.

DETAILED DESCRIPTION:
In this prospective observational trial 7 cohorts of 4 participants each are investigated. The cohorts consist of physicians working at different places in the operating theatre with different occupational exposure to sevoflurane, and one cohort not working in the operating theatre at all. In order to determine the extent of occupational exposure to sevoflurane a human biomonitoring is conducted. Urinary Sevoflurane and its metabolite hexafluoroisopropanol (HFIP) are measured after 3 consecutive working days.

UPDATE: After detecting traces of HFIP in all cohorts even in physicians not working in the operating theatre measurements were repeated, more cohorts were added including a negative control and measurements before the study period of 3 consecutive working days were added.

UPDATE: For comparison one cohort of patients having undergone sevoflurane anaesthesia was added.

ELIGIBILITY:
Inclusion Criteria:

* Occupational exposure to sevoflurane while conducting sevoflurane anaesthesia/being present during sevoflurane anaesthesia
* Possible occupational exposure to sevoflurane while working in the operating room/perioperative anaesthesia care unit
* No occupational exposure to sevoflurane (working outside the operating theatre)

Exclusion Criteria:

* Presence during a mask induction with sevoflurane

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Physicans with or without occupational exposure to sevoflurane.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2021-03-22 (Actual); Study Completion 2021-03-22 (Actual)

PRIMARY OUTCOMES:
Urinary HFIP concentration (µg/l) | After 3 consecutive days of work
  After 3 consecutive days of work a urine sample is collected and urinary HFIP is measured by gas chromatography
Urinary sevoflurane concentration (µg/l) | After 3 consecutive days of work
  After 3 consecutive days of work a urine sample is collected and urinary sevoflurane is measured by gas chromatography

CONTACTS AND LOCATIONS:
Overall Officials: Katharina Roeher, Dr. med, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- Universitätsklinikum Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No